CLINICAL TRIAL: NCT03788031
Title: Towards Developing a Perceptual Learning Treatment for Amblyopia
Brief Title: Perceptual Learning Treatment for Amblyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20171108002
Record Dates: First submitted 2018-12-11; First posted 2018-12-27 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2021-08

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Perceptual learning group - Amblyopia (Experimental): Visual training
  Interventions: Other: Acuity training
- Perceptual learning group - Control (Active Comparator): Visual training
  Interventions: Other: Acuity training
- Occlusion therapy - Amblyopia (Placebo Comparator): Patching
  Interventions: Other: Occlusion therapy

INTERVENTIONS:
Other: Acuity training — The intervention will be a vision therapy. On each trial, a properly oriented stimulus will be presented randomly at one of the four locations on a flat monitor screen. The visual task is to identify the location of the stimulus.
  Arms: Perceptual learning group - Amblyopia; Perceptual learning group - Control
Other: Occlusion therapy — Participants will be required to patch the good eye for 20 days, 1 hour per day.
  Arms: Occlusion therapy - Amblyopia

SUMMARY:
Objectives. To develop a new treatment for amblyopia using a perceptual learning approach.

Hypothesis to be tested. Our proposed experiments are designed to investigate whether practicing a grating detection task can improve vision in patients with amblyopia.

Design and subjects. A total of 36 patients with amblyopia will be randomized allocated into two intervention groups: Group 1, perceptual learning therapy. Group 2, occlusion therapy. A control group comprising of 18 subjects with normal vision will be recruited for comparison. A battery of tests will be used to assess a range of visual functions before and after the treatment intervention.

Study instruments. Grating acuity testing system

Interventions. We have established a clinical protocol for acuity training. On each trial, a properly oriented stimulus will be presented randomly at one of the four locations on a flat monitor screen. The visual task is to indicate the location of the stimulus. Participants will be required to undertake 20 one-hour sessions of training.

Main outcome measures. Resolution acuity, visual acuity, contrast sensitivity function

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity in the amblyopic eye: 20/25 or worse

Exclusion Criteria:

* Manifest eye disease & nystagmus

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change of grating acuity | 20 hours
  Grating acuity tests the participants' ability to resolve fine details. This study measures the change of grating acuity after 20 hours of vision training.

SECONDARY OUTCOMES:
Change of visual acuity | 20 hours
  Visual acuity tests the participants' ability to resolve letters.This study measures the change of visual acuity after 20 hours of vision training.
Change of contrast sensitivity | 20 hours
  Contrast sensitivity reflects the participants' sensitivity to identify low contrast visual stimuli. This study measures the change of contrast sensitivity after 20 hours of vision training.
Change of stereopsis | 20 hours
  Visual acuity tests the 3-D perception. This study measures the change of stereopsis after 20 hours of vision training.

CONTACTS AND LOCATIONS:
Overall Officials: Tsz Wing Leung, Ph.D., Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Optometry Research Clinic, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Levi DM, Li RW. Improving the performance of the amblyopic visual system. Philos Trans R Soc Lond B Biol Sci. 2009 Feb 12;364(1515):399-407. doi: 10.1098/rstb.2008.0203. PMID 19008199
- [Result] Li RW, Klein SA, Levi DM. Prolonged perceptual learning of positional acuity in adult amblyopia: perceptual template retuning dynamics. J Neurosci. 2008 Dec 24;28(52):14223-9. doi: 10.1523/JNEUROSCI.4271-08.2008. PMID 19109504
- [Result] Li RW, Ngo C, Nguyen J, Levi DM. Video-game play induces plasticity in the visual system of adults with amblyopia. PLoS Biol. 2011 Aug;9(8):e1001135. doi: 10.1371/journal.pbio.1001135. Epub 2011 Aug 30. PMID 21912514